CLINICAL TRIAL: NCT01447030
Title: Langtidsopfølgning Efter Kirurgisk Behandling af Iatrogene galdevejslæsioner opstået i Forbindelse Med Cholecystektomi
Brief Title: Long Time Follow up After HJ Following Iatrogenic Bile Duct Injuries
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other); Herlev Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicolaj Markus Stilling, Doctor, Odense University Hospital
Other Study IDs: NMS1
Record Dates: First submitted 2011-10-02; First posted 2011-10-05 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Biliary Strictur After Hepatojejunostomy (HJ); Morbidity and Mortality After and Around HJ
Keywords: Biliary strictur; Hepatojejunostomy; Iatrogenic major bile duct injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction: Bile duct injury (BDI) after cholecystectomy remains a serious complication with major implications for patient outcome. For most major BDIs, the recommended method of repair is a hepaticojejunostomy (HJ). We conducted a retrospective review from 5 Danish hepatobiliary centres aiming to examine the perioperative and the long-term outcome after reconstructive HJ.

ELIGIBILITY:
Inclusion Criteria:

* All patients with iatrogenic Bile duct injury (BDI) after cholecystectomy reconstructed with hepatojejunostomy/choledochojejunostomy.

Exclusion Criteria:

* Patients with non-cholecystectomy-related BDI or with cholecystectomy-related BDI that had been definitively managed by other techniques.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with iatrogenic bile duct injury (BDI) after cholecystectomy reconstructed with hepatojejunostomia. Collecting data from 5 Danish tertiary hepato-biliary centres from january 1995 to may 2009.
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Stricture of HJ | days to years
  Stricture of hepaticojejunostomy after reconstruction